CLINICAL TRIAL: NCT01415050
Title: Multicentered, Randomized Study of Safety and Efficacy of Whole-body Vibration as add-on to Standard Pharmacological Treatment of Osteoporosis in Post-menopausal Women
Brief Title: Safety and Efficacy of Whole-body Vibration as add-on Treatment of Osteoporosis in Post-menopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: X-pert Med GmbH (Industry)
Responsible Party: Dr. med. habil. Matthias Rother, X-pert Med GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPM-022
Record Dates: First submitted 2011-08-01; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis in Post-menopausal Women
Keywords: Osteoporosis; Menopause; Raloxifane; Alendronate
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Active Comparator)
  Interventions: Device: Whole body vibration
- Raloxifane (Active Comparator)
  Interventions: Device: Whole body vibration

INTERVENTIONS:
Device: Whole body vibration — 15 times WBV

SUMMARY:
Multicentered, randomized study of safety and efficacy of whole-body vibration (WBV) as add on to standard pharmacological treatment of osteoporosis (alendronate 70 mg/ week or raloxifene 60 mg/day) in post-menopausal women.

After informed consent of the patients has been obtained, each patient's potential eligibility will be assessed during a "Screening Visit". Eligible subjects will be stratified into two groups: those that are on treatment with alendronate and those that are on treatment with raloxifene.

Subsequently, at baseline, the patients in each group are randomised to receive either WBV or no WBV during the first segment of the study. Baseline evaluation of biomarkers of bone remodelling, fall risk and back pain will be performed before starting the first segment. Patients will return for efficacy and safety evaluations at week 3 and week 6. At 6 weeks after baseline the second segment of the study starts: patients that were on WBV during segment I will be observed for another 6 weeks without WBV, whereas the patients that did not receive WBV during segment I will now be treated with WBV for 6 weeks in segment II. All patients will return for additional visits at week 9 and 12 for safety and efficacy evaluation.

DETAILED DESCRIPTION:
Objectives Primary

1. To establish the effect of whole-body vibration (WBV) on biomarkers of bone remodelling in postmenopausal women with osteoporosis.
2. To establish the effect of whole-body vibration (WBV) on fall risk and low back pain in postmenopausal women with osteoporosis.

Secondary

1. To compare the effects of WBV treatment to the effects of treatment without WBV on biomarkers of bone remodelling, fall risk and low back pain, while keeping standard pharmacotherapy as a constant parameter
2. To compare the effects of WBV in combination with alendronate to the effects of WBV in combination with raloxifene on biomarkers of bone remodelling, fall risk and low back pain
3. To evaluate the long-term effects of WBV on biomarkers of bone remodelling, fall risk and low back pain
4. Safety of WBV

Study Design Multicentered, randomized study of safety and efficacy of whole-body vibration (WBV) as add on to standard pharmacological treatment of osteoporosis (alendronate 70 mg/ week or raloxifene 60 mg/day) in post-menopausal women.

After informed consent of the patients has been obtained, each patient's potential eligibility will be assessed during a "Screening Visit". Eligible subjects will be stratified into two groups: those that are on treatment with alendronate and those that are on treatment with raloxifene.

Subsequently, at baseline, the patients in each group are randomised to receive either WBV or no WBV during the first segment of the study. Baseline evaluation of biomarkers of bone remodelling, fall risk and back pain will be performed before starting the first segment. Patients will return for efficacy and safety evaluations at week 3 and week 6. At 6 weeks after baseline the second segment of the study starts: patients that were on WBV during segment I will be observed for another 6 weeks without WBV, whereas the patients that did not receive WBV during segment I will now be treated with WBV for 6 weeks in segment II. All patients will return for additional visits at week 9 and 12 for safety and efficacy evaluation.

Number of Subjects Total number: 80 patients Group I: Patients on alendronate, n=40 Group I a: WBV in segment I, no WBV in segment II, n= 20 Group I b: no WBV in segment I, WBV in segment II, n=20 Group II: Patients on raloxifene, n=40 Group II a: WBV in segment I, no WBV in segment II, n= 20 Group II b: no WBV in segment I, WBV in segment II, n=20

Diagnosis / Main Inclusion Criteria Ambulatory postmenopausal women, who had their last menstrual period at least 2 years before beginning the study Free of severe acute or chronically disabling conditions with a life expectancy of at least 5 years Expected to remain ambulatory throughout the entire study and expected to return for all study visits Expected to be compliant with study procedures, including procedures for WBV usage Women who have no language barrier, are cooperative, and who give informed consent before entering the study Women must be on standard therapy with alendronate or raloxifene for at least 3 months before the commencement of WBV, and their treatment must be expected to remain stable throughout the study

Main Exclusion Criteria Participation in another clinical study within the last 30 days and/or during the study Subjects who are inmates of psychiatric wards, prisons, or any other state institutions Investigators or any other team member involved directly or indirectly in the conduct of the clinical study Thrombophlebitis, deep venous thrombosis, any thromboembolic disorders (including pulmonary or retinal embolism) within the last year Any vascular disorders of the lower extremities with the exception of asymptomatic varicosis Current bone disorders other than primary osteoporosis, such as hyperparathyroidism, Paget's disease, renal osteodystrophy, osteomalacia, osteonecrosis, spondylolisthesis Vertebral fracture or fractures of the lower extremities within the last 6 months before start of WBV Frequent occurrence of muscle spasms limiting the use of WBV Spastic disorders Morbus Sudeck (CRPS I) Malignancy within the past 2 years with the exception of in situ removal of basal cell carcinoma Severe cardiovascular disorder, such as but not limited to: not controllable hypertension, clinically relevant cardiac arrhythmia and cardiac valve disorder, heart failure (NYHA III-IV) Cerebral vascular accident within the past 1 year Any neurologic/psychiatric disorder which might interfere with the conduct of the trial or the study results such as, but not limited to, the following: Depression, schizophrenia, dementia, Parkinson's disease, epilepsy Benign Paroxysmal Positional Vertigo Frequent occurrence of migraine attacks (more than once per month), limiting the use of WBV Active renal lithiasis or gall stones as defined by any colic within 6 months prior to start of WBV Acute inflammation, infection and/or fever Immune compromised conditions such as, but not limited to, rheumatoid arthritis, HIV severe diabetes, e.g. defined by the coexistence of an arterial occlusive disease Major surgical interventions within 3 months prior to WBV Metallic or plastic implants like joint implants, pace makers, cardiac valves, stents, eye lenses that limit the use of WBV Any acute joint inflammation of the lower extremities or other parts of the body which might interfere with the use of WBV within the last 6 months before start of WBV Start or change in regimen of physical therapy, or extreme sportive activity within 1 month prior to study and during the study Treatment with doses of any of the following medications more recently than 6 months before beginning the study: Androgen, Calcitonin, Estrogen, Progestin, strontium ranelate, parathormone, proton pump inhibitors Long term treatment (more than 6 months) with Heparin within the last 2 years Patients in the alendronate group must be naïve to other bisphosphonates and raloxifen Patients in the raloxifen group must be naïve to all bisphosphonates Treatment with WBV within the last 6 months Treatment with therapeutic doses of systemic corticosteroids for more than 1 month during the 12 months before beginning the study Treatment with 50,000 IU or more of vitamin D once weekly more recently than 3 months before beginning the study

Investigational Medical Device (IMD)

Whole Body Vibration procedure (WBV) will be performed using Fitvibe® medical (Manufacturer: Uniphy Elektromedizin GmbH & Co. KG, Germany), a certified medical device, in the following way:

Three Sessions per week of treatment, with a minimum of 15 sessions within a period of 6 weeks One session consists of 10 runs each containing 30 sec vibration intervals with a 15 sec plateau, interrupted by 30 sec pauses Frequency of 30 Hz Amplitude of 2 mm

Efficacy Endpoints Primary

1. Changes in biomarkers of bone formation (Bone specific alcalic phosphatase - Ostase) and bone resorption (cross links of N-terminal telopeptide of type 1 collagen - N-Tx) during treatment with WBV
2. Changes in fall risk (Tinetti Mobility test) and low back pain (11 point NAS) during treatment with WBV

Secondary

1. Changes in Ostase and N-Tx biomarkers during the first 3 weeks of treatment with WBV
2. Changes in Ostase and N-Tx biomarkers during Segment II in Group I a and II a
3. Changes in fall risk (Tinetti Mobility test) and low back pain (11 point NAS) during the first 3 weeks of treatment with WBV
4. Changes in fall risk (Tinetti Mobility test) and low back pain (11 point NAS) during Segment II in Group I a and II a

Safety Variables Routine physical examinations, monitoring of vital signs, body height and adverse events

Statistical Methods The confirmatory analysis is based on the primary criterion "Effect of WBV", measured with the changes in markers of bone formation Ostase and N-Tx as well as fall risk and low back pain from start to end of WBV segment of the study (within group comparison). Since normal distribution cannot be assumed for the test variables, the Wilcoxon-rank-test will be used as two-sided test on difference.

The final evaluation of the primary criteria will be performed hierarchically in the following order:

1. "changes in marker Ostase during treatment with WBV"
2. "changes in marker N-Tx during treatment with WBV"
3. "changes in fall risk during treatment with WBV"
4. "changes in low back pain during treatment with WBV"

The hypothesis for the four tests on difference are:

H0: µ1-µ2 = 0 H1: µ1-µ2 = 0 The experiment wise multiple level alpha is defined as alpha = 0.05 two-sided respectively as required for confirmatory studies. If the primary hypothesis tests are performed in the given order (1. to 4.) the test can be performed with full alpha as long as the result for the previous test turns to be significant (Principle of a priori ordered hypotheses).

The confirmatory analysis is performed using the ITT population (intention-to-treat).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women, who had their last menstrual period at least 2 years before beginning the study
* Free of severe acute or chronically disabling conditions with a life expectancy of at least 5 years
* Expected to remain ambulatory throughout the entire study and expected to return for all study visits
* Expected to be compliant with study procedures, including procedures for WBV usage
* Women who have no language barrier, are cooperative, and who give informed consent before entering the study
* Women must be on standard therapy with alendronate or raloxifene for at least 3 months before the commencement of WBV, and their treatment must be expected to remain stable throughout the study

Exclusion Criteria:

* Participation in another clinical study within the last 30 days and/or during the study
* Subjects who are inmates of psychiatric wards, prisons, or any other state institutions
* Investigators or any other team member involved directly or indirectly in the conduct of the clinical study
* Thrombophlebitis, deep venous thrombosis, any thromboembolic disorders (including pulmonary or retinal embolism) within the last year
* Any vascular disorders of the lower extremities with the exception of asymptomatic varicosis
* Current bone disorders other than primary osteoporosis, such as hyperparathyroidism, Paget's disease, renal osteodystrophy, osteomalacia, osteonecrosis, spondylolisthesis
* Vertebral fracture or fractures of the lower extremities within the last 6 months before start of WBV
* Frequent occurrence of muscle spasms limiting the use of WBV
* Spastic disorders
* Morbus Sudeck (CRPS I)
* Malignancy within the past 2 years with the exception of in situ removal of basal cell carcinoma
* Severe cardiovascular disorder, such as but not limited to: not controllable hypertension, clinically relevant cardiac arrhythmia and cardiac valve disorder, heart failure (NYHA III-IV)
* Cerebral vascular accident within the past 1 year
* Any neurologic/psychiatric disorder which might interfere with the conduct of the trial or the study results such as, but not limited to, the following: Depression, schizophrenia, dementia, Parkinson's disease, epilepsy
* Benign Paroxysmal Positional Vertigo
* Frequent occurrence of migraine attacks (more than once per month), limiting the use of WBV
* Active renal lithiasis or gall stones as defined by any colic within 6 months prior to start of WBV
* Acute inflammation, infection and/or fever
* Immune compromised conditions such as, but not limited to, rheumatoid arthritis, HIV
* severe diabetes, e.g. defined by the coexistence of an arterial occlusive disease
* Major surgical interventions within 3 months prior to WBV
* Metallic or plastic implants like joint implants, pace makers, cardiac valves, stents, eye lenses that limit the use of WBV
* Any acute joint inflammation of the lower extremities or other parts of the body which might interfere with the use of WBV within the last 6 months before start of WBV
* Start or change in regimen of physical therapy, or extreme sportive activity within 1 month prior to study and during the study
* Treatment with doses of any of the following medications more recently than 6 months before beginning the study: Androgen, Calcitonin, Estrogen, Progestin, strontium ranelate, parathormone, proton pump inhibitors
* Long term treatment (more than 6 months) with Heparin within the last 2 years
* Patients in the alendronate group must be naïve to other bisphosphonates and raloxifen
* Patients in the raloxifen group must be naïve to all bisphosphonates
* Treatment with WBV within the last 6 months
* Treatment with therapeutic doses of systemic corticosteroids for more than 1 month during the 12 months before beginning the study
* Treatment with 50,000 IU or more of vitamin D once weekly more recently than 3 months before beginning the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Biomarkers of bone formation and resorption | 6 weeks
  1. Changes in markers of bone formation (N-terminal propeptide of type-1 procollagen - P1NP) and bone resorption (cross links of N-terminal telopeptide of type 1 collagen - N-Tx) from baseline to week 6

SECONDARY OUTCOMES:
Fall risk | 6 weeks
  Changes in Fall Risk (Tinetti Mobility test) from baseline to week 6
Low back pain | 6 weeks
  Changes in low back pain (100 mm VAS) from baseline to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Egbert Seidel, Prof.Dr.med., Principal Investigator — Zentrum für Physikalische und Rehabilitative Medizin des Sophien- und Hufeland-Klinikums Weimar; Matthias Rother, Dr.med.habil, Study Director — X-pert Med GmbH
Locations (5):
- Germany (5):
  - GP Office Dr. Baumann, Annaberg-Buchholz
  - X-pert Med GmbH, MUC, Gräfelfing
  - X-pert Med GmbH, Jena, Jena
  - Sportmedizin Stockach, Stockach
  - Sophien- und Hufeland- Klinikum GmbH, Weimar